CLINICAL TRIAL: NCT03149770
Title: Hypoglycemia After Exercise in Type 1 Diabetes: Intranasal Naloxone as a Novel Therapy to Preserve Hypoglycemia Counterregulation
Brief Title: Naloxone, Hypoglycemia and Exercise
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MED-2017-25555
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Experimental): Naloxone, then placebo
  Interventions: Drug: Naloxone then placebo
- 2 (Placebo Comparator): Placebo, then Naloxone
  Interventions: Drug: Placebo then Naloxone

INTERVENTIONS:
Drug: Naloxone then placebo — naloxone intranasal 4mg, then placebo
  Arms: 1
Drug: Placebo then Naloxone — placebo then naloxone intranasal 4mg
  Arms: 2

SUMMARY:
The overall objective of this project is to determine if the intranasal administration of naloxone during exercise will be a novel approach to preserve the counterregulatory response to hypoglycemia experienced the next day in patients with type 1 diabetes. Exercise induced autonomic failure contributes to the development of impaired awareness of hypoglycemia. Treatments that blunt the consequences of exercise induced autonomic failure, such as preserving the post-exercise counterregulatory response to hypoglycemia, may improve awareness of hypoglycemia. Naloxone, an opioid antagonist, is an extremely promising agent. In healthy volunteers, intravenous administration of naloxone during exercise preserved the counterregulatory response to hypoglycemia the following day (1). In this study, investigators will extend the clinical applicability by administering intranasal naloxone to individuals with type 1 diabetes. Specifically, the investigators will use a randomized, placebo controlled, crossover design to administer drug or placebo to patients with type 1 diabetes during acute exercise and assess the counterregulatory response to hypoglycemia the following day. The use of intranasal naloxone is a highly innovative aspect of this proposal. Intranasal naloxone translates readily to clinical use and, as demonstrated by the investigators preliminary data, achieves similar plasma drug concentrations as after IV administration.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed on clinical grounds (history of DKA, use of insulin within 6 months of diagnosis)
* Diabetes duration < 30 years (impaired awareness of hypoglycemia increases with duration so it will be more likely that shorter duration participants will have hypoglycemia awareness) but > 2 years (to ensure that they have lost hypoglycemia induced glucagon secretion as is typical in patients who develop impaired awareness of hypoglycemia)
* Age 18 - 65 years
* Baseline hemoglobin A1C 6.8 - 9.0% (range selected to reduce the risk of hypoglycemia and uncontrolled diabetes in the weeks before the study, both of which may affect the responses to hypoglycemia)
* Awareness of hypoglycemia as verified by Cox questionnaire

Exclusion Criteria:

* History of stroke, seizures (other than those related to hypoglycemia), arrhythmias, active cardiac disease
* History of hypertension or blood pressure > 140/95 mm Hg at screening visit
* Pregnancy or plan to become pregnant during the study period
* Health related limitations in exercise (including but not limited to: angina, uncontrolled asthma, peripheral arterial disease)
* Unwillingness to avoid exercise during the 7 days before each part of the study
* Concomitant medical problems that may prevent the participant from successfully completing the protocol
* Smoking as defined by 2 or more tobacco cigarettes a week
* Daily use of opioids or an opioid antagonist or use in the past two weeks
* Unwillingness to wear a continuous glucose monitor for one week before and one week after each part of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Naloxone First, Then Placebo: Naloxone, then placebo
  Naloxone then placebo: naloxone intranasal 4mg, then placebo
- Placebo First, Then Naloxone: Placebo, then Naloxone
  Placebo then Naloxone: placebo then naloxone intranasal 4mg
Period: Overall Study
Arm/Group | Naloxone First, Then Placebo | Placebo First, Then Naloxone
Started | 16 | 14
Completed | 14 | 14
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Naloxone, then placebo
  Naloxone then placebo: naloxone intranasal 4mg, then placebo
- Arm 2: Placebo, then Naloxone
  Placebo then Naloxone: placebo then naloxone intranasal 4mg
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptom Score
Description: The primary outcome variable for Aim 1 will be the difference, naloxone vs. saline, in symptom scores collected using a standard questionnaire during the hypoglycemic clamp on Day 2, after administration of intranasal treatment during exercise on Day 1.
  the scale for symptoms score is 0-72. A higher score represents a better outcome.
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Naloxone: naloxone intranasal 4mg
- Placebo: Participants receiving placebo
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 28 | 26
score on a scale | 25 (12) | 21 (13)

2. Primary Outcome: Change in Epinephrine Levels
Description: The primary outcome variable for Aim 2 will be the difference, naloxone vs. saline, in peak epinephrine levels measured during the hypoglycemic clamp on Day 2, after administration of treatment during exercise on Day 1.
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Placebo: Participants that received placebo
Arm/Group | Naloxone | Placebo
Number analyzed (Participants) | 28 | 26
pg/ml | 425 (236) | 367 (228)

ADVERSE EVENTS:
Time Frame: 3-6 months
Arm/Group | Naloxone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 4/28 | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naloxone (N=28) | Placebo (N=26)
Nausea/vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
headache (General disorders) | 2 (2) | 0 (0)
fatigue/tiredness (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT03149770/Prot_SAP_001.pdf